CLINICAL TRIAL: NCT05409105
Title: Influence of 2-Weeks Mango Ingestion on Inflammation Resolution After Vigorous Exercise
Brief Title: Mangoes and Exercise Inflammation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Appalachian State University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Prevention
Other Study IDs: 22-0127
Record Dates: First submitted 2022-05-12; First posted 2022-06-08 (Actual); Last update posted 2023-06-12 (Actual); Status verified 2023-06

CONDITIONS: Inflammatory Response; Muscular Injury
Keywords: mangoes; exercise; inflammation; oxylipins; inflammasome
MeSH Terms: conditions — Motor Activity; Inflammation | interventions — Water

STUDY DESIGN:
Intervention Model Description: Randomized treatment, crossover
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Mangoes (Experimental): Frozen mangoes, 2 cups per day (with 2 cups water), 2 weeks.
  Interventions: Dietary Supplement: Mangoes
- Water (Active Comparator): Bottled water, 2 cups per day
  Interventions: Dietary Supplement: Water

INTERVENTIONS:
Dietary Supplement: Mangoes — Frozen mangoes, 2 cups per day, 2 weeks
  Arms: Mangoes
Dietary Supplement: Water — 2 cups/day bottled water, 2 weeks
  Arms: Water

SUMMARY:
Vigorous exercise bouts result in significant inflammation and muscle soreness. Our research group has published several papers showing that ingestion of various types of fruits enhances inflammation resolution after exercise. Mangoes have a unique nutrient profile (carotenoids, polyphenols, sugars, vitamins) that we hypothesize will mitigate post-exercise inflammation and muscle soreness. This study will examine the effect of 2 cups/day frozen mango ingestion (2 weeks, 330 g/day) in moderating exercise-induced (2.25 h cycling) inflammation and muscle soreness in a randomized crossover trial. Participants will include 20 male and female young adult cyclists (ages 18-60 years) who are capable of cycling 2.25 h in the laboratory on trainers. In random order, the cyclists will supplement their diets with 2 cups/day mangoes with 1 cup water or 1 cup water alone for two weeks, followed by the 2.25-h exercise challenge. Blood and urine samples will be collected pre- and post-2 weeks supplementation. Additional blood samples will be collected immediately post-exercise, and then 1.5-h, 3-h, and 24-h post-exercise. Urine samples will be analyzed for mango-related metabolites to confirm compliance to the supplementation regimen and to establish statistical relationships with inflammation-related outcomes. The blood samples will be analyzed for novel, cutting-edge outcomes related to inflammation including 70 oxylipins, inflammasome activation, and pro-inflammatory cytokines that we have previously shown are sensitive to exercise and nutrition-based interventions. If the data support our hypothesis, mango ingestion will be viewed as a nutritional strategy to counter exercise-induced inflammation by fitness enthusiasts and athletes who exercise vigorously on a regular basis.

DETAILED DESCRIPTION:
Subjects will come to the lab for orientation/baseline testing, pre-and post-supplementation (2 weeks mango ingestion compared to water alone) blood and urine sample collections with 3-d food records, two 2.25 h cycling sessions, and additional lab visits to provide 1-day 7:00 am recovery blood samples) (thus 7 total lab visits). The total amount of time subjects will be asked to volunteer for this study is about 20 hours at the Human Performance Laboratory (over a 6-week period).

A. Orientation/Baseline Testing (Visit #1):

After voluntarily signed IRB-approved consent forms, study participants will be tested for maximal aerobic capacity (VO2max) during a graded, cycling test with continuous metabolic monitoring with the Cosmed CPET metabolic device (Cosmed, Rome, Italy). Body composition will be measured with the seca BIA and Bod Pod body composition analyzer (Life Measurement, Concord, CA). Demographic and training histories will be acquired with questionnaires. A symptom inventory will be conducted using a 2-week retrospective questionnaire. 3-day food records and 24-h urine collection kits will be supplied with thorough instructions.

B. Pre-Supplementation Lab Visit #2 and 2-Week Mango Supplementation Protocol:

Two weeks prior to the first running session, subjects will report to the Human Performance Laboratory at approximately 7:00-8:00 am. A blood sample will be collected in an overnight fasted state to coincide with the same time of the day for the post-supplementation blood draw. Urine samples and 3-d food records will be turned in after review. A 2-week supply of frozen mangoes in date/time labeled freezer bags (1 cup or 165-gram amounts) will be given to the participants randomized to the mango trial, with instructions to consume 1 cup each with the first and last meals of the day (for two weeks). Participants will be given the frozen mangoes in cold containers and then instructed to store these in their home freezers. Subjects will be instructed to consume the mangoes in a variety of ways including in smoothies, with yogurt, or as is. Bottled water will be supplied to both groups with instructions to consume 1 cup each with the first and last meals of the day. Subjects will be instructed to store and then bring the freezer bags to their next lab visit. To assess potential adverse effects, a symptom inventory will be conducted using a 2-week retrospective questionnaire (before and after the 2-week supplementation period). Rationale for the mango dosing regimen: The amounts of carotenoids and polyphenols in 2 cups/d mangoes are similar to amounts we have used successfully in prior studies to mitigate post-exercise inflammation and muscle soreness. We recommend a 2-week supplementation period because our experience is that this is a sufficient time period for bioactive effects to emerge as the gut microbiome and tissues adapt. We recommend using water as the control condition to allow the full array of nutrient components found in mangoes (carbohydrate, carotenoids, polyphenols, vitamins C and A) to be tested when compared to just water.

C. 2.25 h Cycling Session (Lab Visit #3):

During the 3-day period prior to the 2.25-h cycling session, subjects will taper exercise training and ingest a moderate-carbohydrate diet using a food list restricting high fat foods, visible fats, and polyphenols. Subjects will record all food and beverage intake during the 3-day period, with macro- and micro-nutrient intake assessed using the Food Processor dietary analysis software system (ESHA Research, Salem, OR). We will also measure total flavonoid intake (and 6 flavonoid subgroups) using the USDA flavonoid database that we have incorporated into the Food Processor database. Study participants will report to the Human Performance Lab in an overnight fasted state and provide a blood sample, ingest 1 cup mango with 1 cup of water, or 1 cup of water alone, and then cycle 2.25 h at high intensity (70% VO2max) while ingesting water alone (3 ml/kg every 15 minutes). Blood samples will be collected at 0 h, 1.5 h, 3.0 h, and 24 h post-exercise.

Testing protocol during the lab sessions with the 2.25-h cycling session:

1. 7:00 am: Provide blood sample, delayed onset of muscle soreness (DOMS) rating (1-10 scale), profile of mood states ratings (POMS), and turn in the 24-h urine sample and 3-day food record. Fill in the 2-week retrospective symptom log.
2. 7:10 am: Ingest 1 cup mangoes with 1 cup water or 1 cup water alone.
3. 7:30 am: Start the 2.25 h cycling session. Subjects will cycle on trainers in the lab at 70% VO2max (~race pace) for 2.25 hours. Oxygen consumption, carbon dioxide production, respiratory exchange ratio, and ventilation will be measured using the Cosmed Quark CPET metabolic cart after 15 minutes and then every 30 minutes. Subjects will consume 3 ml/kg water every 15 min. No other beverage or food containing energy or nutrients will be allowed during the 2.25-h cycling sessions.
4. ~10:00 am to 1:00 pm: Blood samples will be taken via venipuncture immediately after completing the cycling session, and then 1.5-h and 3.0-h post-exercise. Subjects will be allowed to shower and change clothes. The DOMS and POMS questionnaires will be administered each time blood samples are collected. Subjects will ingest no food or beverage other than water (7 ml/kg during the 1.5 h post-exercise period). After the 1.5 h post-exercise blood draw, subjects in the mango group will consume 1 cup mangoes with 1 cup of water. Subjects in the water group will consume a calorie-matched volume of Gatorade (0.45 liters). Another blood sample will be collected 3-h post-exercise. Afterwards, subjects will be allowed to leave the lab with instructions to adhere to the food list requirements, and to keep exercise training moderate.
5. 7:00 am, next morning: 24-h blood sample and DOMS and POMS ratings (Lab visit #4).

D. Washout/Crossover/Repeat Subjects will engage in a 2-week washout period without the mango supplements, crossover to the opposite treatment arm, and then repeat all procedures (Lab visits #5,6,7).

ELIGIBILITY:
Inclusion Criteria:

* Male or female cyclist, ages 18-60 years, and capable of cycling 2.25 h in the lab on trainers at 70% VO2max (close to race pace).
* Non-smoker, and generally healthy and without chronic disease including cardiovascular disease (e.g., heart disease, stroke), cancer, type 1 and 2 diabetes, rheumatoid arthritis. Categorized as "low risk" using the American College of Sports Medicine screening questionnaire.
* Agree to train normally, maintain weight, and avoid the regular use of large-dose vitamin and mineral supplements, herbs, and medications that influence inflammation (especially NSAIDs) for the duration of the 6-week study and at least a 2-week period prior to the study.
* Agree to taper their exercise routine prior to each of the two lab cycling sessions.
* Agree to avoid ingestion of mangoes (fresh or within other products) during the study (other than provided).

Exclusion Criteria:

* Inability to comply with study requirements, history of allergic reactions to mangoes.
* Females: body weight below 110 pounds; pregnant or breastfeeding.
* Any other concurrent condition which, in the opinion of the principle investigator (PI), would preclude participation in this study or interfere with compliance.
* Current diagnosis of cardiovascular disease, diabetes, or cancer (except for non-melanoma skin cancer).

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 22 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-12-31 (Actual); Study Completion 2023-01-30 (Actual)

PRIMARY OUTCOMES:
Plasma lipid mediators | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Plasma concentrations of arachadonic acid oxidized derivatives from LC-MS-MS analysis

SECONDARY OUTCOMES:
Urine mango metabolites | Change from pre-study to post-2 weeks supplementation
  Urine mango polyphenol metabolites
Plasma inflammasome activation | Change from pre-study to post-2 weeks supplementation, and immediately post-exercise, and 1.5 hours-, 3 hours-, and 24 hours-post-exercise
  Plasma concentrations of ASC oligomers from ELISA analysis

CONTACTS AND LOCATIONS:
Overall Officials: David C Nieman, DrPH, Principal Investigator — Appalachian State Univ
Locations (1):
- Appalachian State University Human Performance Lab, North Carolina Research Campus, Kannapolis, North Carolina, United States

IPD SHARING:
Plan to Share IPD: Yes
Will share data upon request.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: December 2022, indefinitely
Access Criteria: Upon request.